CLINICAL TRIAL: NCT06703450
Title: Noninvasive Diagnosis of Liver Fibrosis With Gadopiclenol DCE-MRI in Metabolic Dysfunction-associated Steatohepatitis (MASH)
Brief Title: Guerbet Liver Fibrosis
Status: Enrolling by invitation | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Guerbet (Industry)
Responsible Party: Principal Investigator, Sara Lewis, Radiology Physician, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 23-0855
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2024-11

CONDITIONS: Metabolic Dysfunction-associated Steatotic Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with liver disease: Participants with liver disease for diagnosis of liver fibrosis to have DCE-MRI

SUMMARY:
The goal of this study is to assess the value of liver dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) and texture analysis post gadopiclenol for liver fibrosis staging, in comparison with MR elastography, T1 mapping, ultrasound elastography and blood tests in 50 initial patients with metabolic dysfunction-associated steatohepatitis (MASH).

DETAILED DESCRIPTION:
Metabolic dysfunction-associated steatotic liver disease (MASLD, formerly known as nonalcoholic fatty liver disease or NAFLD) is characterized by the accumulation of excess fat in the liver, ranging from mild forms like non-alcoholic fatty liver (NAFL) to more severe stages such as metabolic dysfunction-associated steatohepatitis (MASH, formerly known as nonalcoholic steatohepatitis or NASH) with associated inflammation, ballooning, fibrosis, and cirrhosis. The severity of MASH and increasing fibrosis stages is associated with higher morbidity and mortality rates. The study will compare dynamic contrast-enhanced (DCE)-MRI measurements of perfusion using gadopiclenol for diagnosis of liver fibrosis to MR elastography and transient elastography, T1 mapping, ultrasound elastography and blood tests, using histopathology as the reference in patients with MASH. In this study, the value of DCE-MRI and texture analysis using gadopiclenol, a new macrocyclic, non-ionic, extracellular contrast agent with high relaxivity will also be assessed which provides, at a lower dose, better contrast-to-noise ratio than gadoterate, gadobenate, and gadobutrol.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected MASLD (F0-F4) with clinically indicated percutaneous or transjugular liver biopsy within 6 months of MRI (before or after MRI).
* Both genders.
* Age > 18 years.
* Any racial/ethnic background.

Exclusion criteria:

* Previous history or current diagnosis of HCC or decompensation.
* Contraindications for MRI, including

  * Medically unstable
  * Intracranial clips
  * Metal implants
  * Suspected or confirmed metal in eyes
  * Cardiac pacemaker, implanted defibrillator, other implanted electronic device
  * Pregnancy: Pregnancy tests will be offered to women of childbearing age at no cost
  * Severe claustrophobia

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing MRI for management of chronic liver disease, such as MASH/NAFLD
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Liver Stiffness by MR Elastography | during procedure (MRI)
  Liver stiffness that is quantitively measured by MR Elastography and correlated with grade of tissue fibrosis from histopathology. Min and Max Scale: 0-20 kilopascals (continuous variable). Higher score indicates poorer health outcomes.

SECONDARY OUTCOMES:
Total Liver Flow | during procedure (MRI)
  Liver Perfusion (DCE MRI) to measure Total liver flow (continuous variable) Max and Min: 0-500 mL/minute per 100g tissue
Arterial Fraction of flow | during procedure (MRI)
  Arterial Fraction of flow - measures and compares the blood flow on both sides of a blockage in the heart's coronary artery to see how much the blockage is affecting blood flow.
Portal Venous Fraction of flow | during procedure (MRI)
  Portal Venous Fraction of flow - measures and compares the blood flow on both sides of a blockage in the heart's coronary artery to see how much the blockage is affecting blood flow.
Distribution volume of contrast | during procedure (MRI)
  Distribution volume of contrast agent

CONTACTS AND LOCATIONS:
Overall Officials: Sara Lewis, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No